CLINICAL TRIAL: NCT01836926
Title: Transanal Minimally Invasive TME (TaTME) Versus Open Intersphincteric Resection and Total Mesorectal Excision of Stage II/III Ultralow Rectal Cancer After Neoadjuvant Concurrent Chemoradiotherapy.
Brief Title: TaTME Versus Open Intersphincteric Resection After Neoadjuvant Concurrent Chemoradiotherapy.
Acronym: TaTME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osama Mohammad Ali ElDamshety (Other)
Collaborators: Mansoura University (Other); Marche Polytechnic university, Ancona, Italy (Unknown)
Responsible Party: Sponsor-Investigator, Osama Mohammad Ali ElDamshety, oncology surgeon--Oncology Centre of Mansoura University (OCMU), Mansoura University
Organization: Mansoura University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mansoura oncology centre
Record Dates: First submitted 2013-04-04; First posted 2013-04-22 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Rectal Cancer
Keywords: sphincter sparing procedures; intersphincteric resection; rectal cancer; ultralow rectal cancer; sphincter preserving procedures; Abdominoperineal resection; Trans-anal minimally invasive surgery; TAMIS versus open colorectal resection; neoadjuvant chemo-radiotherapy for rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open intersphincteric resection (Active Comparator): surgical Instruments for open approach intervention: Open laparotomy through abdominal incision and mobilization of the colon and rectum up to the splenic flexure with high ligation of the inferior mesenteric vessels and mesorectal excision till the levator ani then the peranal approach to resect the distal margin of the rectum through high or low intersphincteric resection in the plane between internal and external anal sphincters.
  Interventions: Procedure: Open intersphincteric resection
- laparoscopic intersphincteric resection . (Active Comparator): instruments used: 4 or 5 laparoscopic trocars (two or three (10-mm) trocar, Two 5-mm trocars and a 12-mm trocar with reducers),Three 5-mm fenestrated grasping forceps, Five-millimetre coagulating shears, a 5-mm straight grasping forceps, Harmonic scalpel, 5 or 10 mm, a 10-mm fenestrated forceps, a 10-mm dissector,5 mm Bipolar grasper, a 5-mm needle holder, Twelve-millimetre linear staplers
  intervention:
  1. Trocar Placement and Exposure
  2. Rectosigmoid Mobilization and Control of Inferior Mesenteric Vessels
  3. Taking Down the Splenic Flexure
  4. rectal dissection till the levator ani muscle and resection of thye lateral ligaments
  then the peranal phase as in the laparotomy approach.
  Interventions: Device: transanal minimally invasive intersphincteric resection

INTERVENTIONS:
Procedure: Open intersphincteric resection — laparotomy arm: surgical Instruments for open approach operation: Abdominal anterior resection combined with peranal intersphincteric resection of the rectum
  Abdominal step a high ligation of the inferior mesenteric artery is performed together with a full mobilization of the left colon. A circular incision of the anal canal is performed 1 cm below the tumour. Both the mucosa and the muscular layer are incised to transect the internal anal sphincter. A coloanal anastomosis, transverse coloplasty or colonic J-pouch and a diverting loop ileostomy are associated with the hand-sewn coloanal anastomosis.
  laparoscopic approach group: instruments used: laparoscopic instruments mentioned at the arm description
  intervention: laparoscopic mobilization of the rectum and colon combined with the peranal intersphincteric resection as in the laparotomy approach
  Other Names: sphincter preserving procedures in low rectal cancer; very low rectal cancer resection; interspincteric resection
  Arms: Open intersphincteric resection
Device: transanal minimally invasive intersphincteric resection — minimally invasive approach group: instruments used: laparoscopic instruments mentioned at the arm description instruments: laparoscopic instruments mentioned in the laparoscopic rectal resection arm intervention: laparoscopic mobilization of the rectum and colon combined with the peranal intersphincteric resection as in the laparotomy approach
  Other Names: laparoscopic low anterior resection combined with trans-anal endoscopic intersphincteric resection; lTAMIS
  Arms: laparoscopic intersphincteric resection .

SUMMARY:
The two surgical options for lower 1/3 rectal cancer is APR and sphincter sparing procedures. Intersphincteric resection is procedure to treat very low rectal cancer within 2 cm from the dentate line to avoid permanent colostomy,improves the quality of life with better genitourinary function. Neoadjuvant chemo-radiotherapy is routine for T3 cases.

DETAILED DESCRIPTION:
During the period between April 2013 and July 2019, a non-randomized controlled study was performed at two tertiary centers; Oncology Centre of Mansoura University and Policlinico Umberto Primo surgery department of SAPIENZA university of Rome after referral from the clinical oncology and nuclear medicine department. After diagnosis of ultralow rectal cancer, a written informed consent was obtained from patients after full explanation of the procedure, the likely outcome and the potential complications that may occur. Digital rectal examination was conducted to assess the distance of lower tumor margin from the anal verge and the anal tone. Anesthetic fitness and tumour markers (CEA) were assessed. Pelvis MRI and/or endorectal ultrasound (EUS), abdomen and chest CT scan and colonoscopy with biopsy were done for all cases. Re-evaluation after neoadjuvant chemo-radiotherapy by MRI and EUS. Inclusion criteria included a very low rectal cancer below 5 cm from the anal verge with normally continent and tumor-free external anal sphincter. Neoadjuvant treatment was given to all patients with T3 or node positive tumors. Exclusion criteria were T4, metastatic tumors and fecal incontinence. Fifty patients were excluded from the study (Fig.1). One hundred and ten patients with ultralow rectal adenocarcinoma, with matched age and sex (table 1), were non-randomly classified into two equal groups: the control group included 55 patents that underwent sphincter sparing by open ISR with TME (O-ISR Group) and the 2nd group included 55 patents that underwent Transanal minimally invasive ISR with TME (TAMIS Group).

Surgical technique:

In open ISR, the inferior mesenteric vessels were highly ligated. After full mobilization of the left colon and splenic flexure was done, the plane for TME was followed down in the pelvis superficial to the hypogastric fascia as low as possible to enter into the posterior intersphincteric plane. A non-endoscopic perineal phase was then initiated using an anal lone-star retractor to expose the anal canal. Both the mucosa and the muscular layer were incised 1cm below the tumor margin to transect the internal anal sphincter (IAS) and then closed by purse string sutures. The dissection continued between IAS and the external anal sphincter (EAS) starting posteriorly then laterally, where EAS is easier to identify, then anteriorly where the plane presented more adhesions with the urethra in male or vagina in female till reaching the abdominal dissection. Proximal division of the specimen started just below the site of inferior mesenteric vessels ligation and continued till division of the marginal artery at the site of the required anastomosis. The Specimen extraction and division was done extra-anal. A defunctioning ileostomy was done in all cases.

In TAMIS-TME, using a lone star retractor, the 1st step was to divide and close the anal canal by purse-string suturing to enter the intersphincteric plane. Using TEo platform (Karl Storz, Tuttilingen, Germany) (fig. 2) with a 4 cm size operating proctoscope diameter, Transanal endoscopic dissection was initiated and continued in the intersphincteric plane starting posteriorly then laterally. Partial or high ISR started at the dentate line to remove the upper half of IAS for ultralow tumors at 3 to 4.5 from anal verge. Total or low ISR started 1 cm below the dentate line, removing the whole of IAS for tumours below 3 cm from the anal verge. The endoscopic dissection continued in the same sequence as the control group along the levator ani. Then continue posteriorly till reaching as much as possible, then dissection continued laterally and anteriorly to reach the peritoneal reflection. Then, the laparoscopic phase was initiated to ligate the inferior mesenteric vessels and mobilize the splenic flexure and left colon. The peritoneal reflections were then divided to connect to the transanal part. The specimen was then extracted transanally and the Colo-anal anastomosis was done in two layers. A defunctioning ileostomy was done in all cases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low rectal carcinoma(The lowest margin of tumor located 3 cm from anal verge ; ≤ 2 cm from dentate lines; 1 cm from anorectal rings.
* Local spread restricted to the rectal wall or the internal anal sphincter.
* Adequate preoperative sphincter function and continence.
* Absence of distant metastasis.

Exclusion Criteria:

* Contraindications to major surgery and American Society of Anesthesiologists (ASA) Physical Status scoring 4.
* Metastatic rectal cancer.
* Those in Dukes stage D (T4 lesion).
* Undifferentiated tumours.
* Local infiltration of external anal sphincter or levator ani muscles.
* Tumor located more than 2 cm above the dentate line.
* Presence of fecal incontinence.
* Patients unwilling to take part in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Early Complications number | 2 years

SECONDARY OUTCOMES:
Duration of the intervention | 1 day
  Duration of surgery
Amount of blood loss and rate of blood transfusion | 1 Day
  Amount of blood loss and blood transfusion through the operation
conversion rate for open ISR | 1 day
The onset of intestinal motility. | 2 weeks
  the onset of the intestinal motility guided by (the onset of borborygmus and its sequence, time to give off flatus, time to intake liquid and solid food)
Pain score | the first two weeks in the postoperative period
  Recording of the needed analgesia guided by pain score
Postoperative hospital stay | 30 Days
  Outcome observers will assess the hospital stay days after both procedures
30 days follow up for re-operation in the postoperative period | 1 month
  readmission within 30 days after patient discharge
Late complications | 2 years
Local recurrence within 2 years | 2 years
  The patients will be observed after the operation for 2 years for local pelvic recurrence
Distant metastasis within 2 years | 2 years
  Distant metastasis after the opertaion for 2 years
Clinical functional outcome | 1 year
  Investigators will assess the continence using Per Anal Scoring System (PASS) from 0 to 4

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mansoura oncology centre, Al Mansurah, Dakahlia Governorate
  - Mansoura university oncology centre, Al Mansurah, Dakahlia Governorate

REFERENCES:
- [Result] [1] Zeeneldin A, Saber M, Seif El-din I, Frag S. Colorectal carcinoma in Gharbiah district, Egypt: Comparison between the elderly and non-elderly. Journal of Solid Tumors 2012; Vol. 2, No. 3. [2] Heald RJ, Husband EM, Ryall RD The mesorectum in rectal cancer surgery-the clue to pelvic recurrence? Br J Surg 1982; 69:613-616 [3] Daniels IR, Fisher SE, Heald RJ, Moran BJ. Accurate staging, selective preoperative therapy and optimal surgery improves outcome in rectal cancer: a review of the recent evidence. Colorectal Dis 2007; 9: 290-301. [4] Sebag-Montefiore D, Stephens RJ, Steele R, Monson J, Grieve R, Khanna S et al. Preoperative radiotherapy versus selective postoperative chemoradiotherapy in patients with rectal cancer (MRC CR07 and NCIC-CTG C016): a multicentre, randomised trial. Lancet 2009; 373: 811-820. [5] Bai X., Li S., Yu B., Su H., Jin W., Chen G., Du J. And Zuo F. Sphincter-preserving surgery after preoperative radiochemotherapy for T3 low rectal cancers. Oncology Letters 2012; 3: 1336-1340 [6] Tytherleigh MG and Mortensen MN. Options for sphincter preservation in surgery for low rectal cancer , British Journal of Surgery 2003; 90: 922-933 DOI: 10.1002/bjs.4296 [7] Schiessel R, Karner-Hanusch J, Herbst F, Teleky B, Wunderlich M. Intersphincteric resection for low rectal tumours. Br J Surg 1994; 81: 1376-1378. [8] Kapiteijn E, Marijnen CA, Nagtegaal ID et al Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer. N Engl J Med 2001; 345:638-646